CLINICAL TRIAL: NCT05220527
Title: Therapeutic Effects of Knee Intra-articular Injections on Patients With Knee Osteoarthritis: a Double-blind, Randomized, Placebo-controlled Clinical Trial
Brief Title: Effects of Knee Injections on Patients With Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MOST109-2314-B-341-001
Record Dates: First submitted 2022-01-05; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Knee Osteoarthritis; Injection; Effect of Drug
Keywords: knee osteoarthritis; steroid; hyaluronic acid; dextrose
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Triamcinolone; Adrenal Cortex Hormones; Hyaluronic Acid; Glucose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study group (Experimental): triamcinolone plus hyruan injection
  Interventions: Drug: Triamcinolone plus hyruan
- Experimental (Active Comparator): vitagen plus hyruan injection
  Interventions: Drug: vitagen plus hyruan
- Placebo (Placebo Comparator): normal saline plus hyruan injection
  Interventions: Drug: normal saline plus hyruan

INTERVENTIONS:
Drug: Triamcinolone plus hyruan — triamcinolone plus hyruan injections, one time per week, for 3 weeks
  Other Names: corticosteroids plus hyaluronic acid
  Arms: Study group
Drug: vitagen plus hyruan — vitagen plus hyruan injections, one time per week, for 3 weeks
  Other Names: dextrose plus hyaluronic acid
  Arms: Experimental
Drug: normal saline plus hyruan — normal saline plus hyruan injections, one time per week, for 3 weeks
  Other Names: normal saline plus hyaluronic acid
  Arms: Placebo

SUMMARY:
Using a double-blind, randomized, placebo-controlled design to compare the immediate, short-term, and intermediate-term additional therapeutic effects of ultrasound-guided corticosteroid injection and dextrose injection to hyaluronic acid injection on patients with knee osteoarthritis, under the basis of International Classification of Functioning, Disability and Health.

DETAILED DESCRIPTION:
A total of 60 patients will be collected. The participants will be randomized into three groups, including the hyaluronic acid combined corticosteroid group, hyaluronic acid combined dextrose group, and hyaluronic acid combined normal saline group (placebo group). The functional performance and knee-related quality of life (Western Ontario and McMaster Universities Osteoarthritis index、Knee Injury and Osteoarthritis Outcome Score), pain (pressure threshold by pain pressure ergometer), and physical activity (10 meters normal and fast walk, up and downstairs, 5 repeated chair-rising time, timed up and go test) and image progression by high-resolution ultrasound will be evaluated before treatment, one week after injections, one month after injections, three months after injections, and six months after injections.

Participants and evaluators will be both blinded to the group's allocation during the whole course of intervention.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of knee osteoarthritis
2. can walk for 15 meters
3. Kellgren-Lawrence grade 2 or greater
4. can follow up for 6 months

Exclusion Criteria:

1. Major diseases will affect balance, such as stroke
2. infectious disease,
3. rheumatoid arthritis,
4. malignancy
5. pregnancy or prepare to pregnant
6. received knee injections in the past 6 months
7. previous knee operation history

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis index | changes of scores from baseline to at one week, one month, 3 months, and 6 months after 3 times of injections
  assess knee related performance, scores: 0-100, higher score indicates a worse outcome

SECONDARY OUTCOMES:
physical functional performance-walking | changes of time (seconds) from baseline to at one week, one month, 3 months, and 6 months after 3 times of injections
  10 meters normal and fast walking speed
physical functional performance-stairs climbing | changes of time (seconds) from baseline to at one week, one month, 3 months, and 6 months after 3 times of injections
  time for up and down stairs
physical functional performance-chair rising | changes of time (seconds) from baseline to at one week, one month, 3 months, and 6 months after 3 times of injections
  time for 5 repeated chair-rising time
physical functional performance-balance | changes of time (seconds) from baseline to at one week, one month, 3 months, and 6 months after 3 times of injections
  time for up and go test
Knee Injury and Osteoarthritis Outcome Score | changes of scores from baseline to at one week, one month, 3 months, and 6 months after 3 times of injections
  assess knee osteoarthritis related function, scores: 0-100, higher score indicates a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Study Chair — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
By request, the data will be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after publication and for one year since publication.
Access Criteria: Request by mail to the investigator.